CLINICAL TRIAL: NCT02927613
Title: Patient Characteristics, Feasibility, and Outcomes of a Home Mechanical Ventilation Program in a Developing Country
Status: Completed | Type: Observational
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Narongkorn Saiphoklang, MD, Assistant Professor, Thammasat University
Other Study IDs: MTU-EC-IM-6-146/57
Record Dates: First submitted 2016-09-30; First posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Home Mechanical Ventilation; Prolonged Mechanical Ventilation
Keywords: Home mechanical ventilation; Mortality; Complications; Developing country

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims to describe the patient characteristics, feasibility, and outcomes of an home mechanical ventilation (HMV) program at a university hospital in Thailand.

DETAILED DESCRIPTION:
Data will be collected on all patients who were discharged with HMV between October 2014 and August 2015 at Thammasat University Hospital. Data include sex, age, co-morbid diseases, clinical features, causes of HMV, mechanical ventilator and complimentary equipment characteristics, caregiver characteristics, ventilator and patient care costs, and morbidity and mortality outcomes of patients.

ELIGIBILITY:
Inclusion Criteria:

* All hospitalized patients requiring mechanical ventilation aged 18 or more years.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All hospitalized patients requiring mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Mortality rate of HMV patients | Up to 1 year
  The number of deaths among HMV patients is recorded during follow-up period (up to 1 year)

SECONDARY OUTCOMES:
Healthcare home visit | Up to 1 year
  Record the number of healthcare home visits (events)
Caregiver characteristics | Up to 1 year
  Record the number of caregivers per patient, the number of well-trained caregivers
Family characteristics | Upto 1 year
  Record types (relationships) and the number of family members, income to costs ratio
HMV complications due to tracheobronchitis | Up to 1 year
  Record the number of tracheobronchitis (events) and the number of hospitalizations due to their effects
HMV complications due to ventilator-associated pneumonia | Up to 1 year
  Record the number of ventilator-associated pneumonias (events) and the number of hospitalizations due to their effects
HMV complications due to the loose tracheostomy | Up to 1 year
  Record the number of loose tracheostomies (events) and the number of hospitalizations due to their effects
HMV complications due to the granulation-tissue formation at tracheostomy | Up to 1 year
  Record the number of granulation-tissue formations at tracheostomy (events) and the number of hospitalizations due to their effects
HMV complications due to pneumothorax | Up to 1 year
  Record the number of pneumothoraces (events) and the number of hospitalizations due to their effects
HMV complications due to the ventilator malfunction | Up to 1 year
  The number of ventilator malfunctions (events) and the number of hospitalizations due to their effects

CONTACTS AND LOCATIONS:
Overall Officials: Narongkorn Saiphoklang, MD, Principal Investigator — Faculty of Medicine, Thammasat University
Locations (1):
- Department of Medicine, Faculty of Medicine, Thammasat University, Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Oktem S, Ersu R, Uyan ZS, Cakir E, Karakoc F, Karadag B, Kiyan G, Dagli E. Home ventilation for children with chronic respiratory failure in Istanbul. Respiration. 2008;76(1):76-81. doi: 10.1159/000110801. Epub 2007 Nov 6. PMID 17984626
- [Background] Divo MJ, Murray S, Cortopassi F, Celli BR. Prolonged mechanical ventilation in Massachusetts: the 2006 prevalence survey. Respir Care. 2010 Dec;55(12):1693-8. PMID 21122178
- [Background] MacIntyre NR, Epstein SK, Carson S, Scheinhorn D, Christopher K, Muldoon S; National Association for Medical Direction of Respiratory Care. Management of patients requiring prolonged mechanical ventilation: report of a NAMDRC consensus conference. Chest. 2005 Dec;128(6):3937-54. doi: 10.1378/chest.128.6.3937. PMID 16354866
- [Background] Kurek CJ, Cohen IL, Lambrinos J, Minatoya K, Booth FV, Chalfin DB. Clinical and economic outcome of patients undergoing tracheostomy for prolonged mechanical ventilation in New York state during 1993: analysis of 6,353 cases under diagnosis-related group 483. Crit Care Med. 1997 Jun;25(6):983-8. doi: 10.1097/00003246-199706000-00015. PMID 9201051
- [Background] Lone NI, Walsh TS. Prolonged mechanical ventilation in critically ill patients: epidemiology, outcomes and modelling the potential cost consequences of establishing a regional weaning unit. Crit Care. 2011;15(2):R102. doi: 10.1186/cc10117. Epub 2011 Mar 27. PMID 21439086
- [Background] McKim DA, Road J, Avendano M, Abdool S, Cote F, Duguid N, Fraser J, Maltais F, Morrison DL, O'Connell C, Petrof BJ, Rimmer K, Skomro R; Canadian Thoracic Society Home Mechanical Ventilation Committee. Home mechanical ventilation: a Canadian Thoracic Society clinical practice guideline. Can Respir J. 2011 Jul-Aug;18(4):197-215. doi: 10.1155/2011/139769. PMID 22059178
- [Background] Sanjuan-Lopez P, Valino-Lopez P, Ricoy-Gabaldon J, Verea-Hernando H. Amyotrophic lateral sclerosis: impact of pulmonary follow-up and mechanical ventilation on survival. A study of 114 cases. Arch Bronconeumol. 2014 Dec;50(12):509-13. doi: 10.1016/j.arbres.2014.04.010. Epub 2014 Jun 12. English, Spanish. PMID 24931271
- [Background] Tagami M, Kimura F, Nakajima H, Ishida S, Fujiwara S, Doi Y, Hosokawa T, Yamane K, Unoda K, Hirose T, Tani H, Ota S, Ito T, Sugino M, Shinoda K, Hanafusa T. Tracheostomy and invasive ventilation in Japanese ALS patients: decision-making and survival analysis: 1990-2010. J Neurol Sci. 2014 Sep 15;344(1-2):158-64. doi: 10.1016/j.jns.2014.06.047. Epub 2014 Jul 1. PMID 25017882
- [Background] Heinemann F, Budweiser S, Jorres RA, Arzt M, Rosch F, Kollert F, Pfeifer M. The role of non-invasive home mechanical ventilation in patients with chronic obstructive pulmonary disease requiring prolonged weaning. Respirology. 2011 Nov;16(8):1273-80. doi: 10.1111/j.1440-1843.2011.02054.x. PMID 21883681
- [Background] Hazenberg A, Kerstjens HA, Prins SC, Vermeulen KM, Wijkstra PJ. Initiation of home mechanical ventilation at home: a randomised controlled trial of efficacy, feasibility and costs. Respir Med. 2014 Sep;108(9):1387-95. doi: 10.1016/j.rmed.2014.07.008. Epub 2014 Jul 22. PMID 25081652
- [Background] Simonds AK. Risk management of the home ventilator dependent patient. Thorax. 2006 May;61(5):369-71. doi: 10.1136/thx.2005.055566. PMID 16648349